CLINICAL TRIAL: NCT00554125
Title: A Prospective Randomised, Open-Labeled Study Comparing Sirolimus Versus FK506 In OLT for Patients With HCC Exceeding Milan Criteria
Brief Title: Sirolimus-Based Immunosuppression Therapy in OLT for Patients With HCC Exceeding Milan Criteria
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZSH-LCI-FJ-0002
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Sirolimus; Orthotopic liver transplantation; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2, III ,intervention (Active Comparator)
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — given at an initial dose of 3 mg/m2, and adjusted over time to achieve steady-state whole-blood trough levels of approximately 5-8 ng/mL

SUMMARY:
The purpose of this study is to evaluate the influence of sirolimus on outcome after OLT for HCC exceeding Milan criteria.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most prevalent cancers in Asia and Africa. Although the first-line therapy for HCC is liver resection, the concomitant cirrhosis often leaves orthotopic liver transplantation (OLT) rather than liver resection as the only potentially curative option. The risk of recurrence is the major concern in patients transplanted for HCC. It has been demonstrated that utilizing more restrictive selection criteria before submitting cirrhotic patients with HCC to liver transplantation is associated with a better outcome. The Milan criteria (one nodule ≤5 cm or 2-3 nodules all <3 cm, without macroscopic vascular invasion and extrahepatic spreading)provide a simple means of selecting patients with HCC for transplantation with a low risk (≈10%) for recurrence. However, the benefit of OLT for patients with HCC within the Milan criteria is opposed by a critical organ shortage, which lengthens the waiting time and thus allows tumor progression during the waiting period. Nearly one third of patients who have a transplant for HCC fall outside the Milan criteria on the basis of pathological findings in the explanted liver, and had a higher risk of tumor recurrence.This led to a dramatic decline in overall and disease-free survival, from 71-85% to 40-50%, and from 65-78% to 27-30%, respectively.

Although it can be hypothesized that the pharmacologic immunosuppression required after liver transplantation for HCC may be accelerated tumor recurrence and metastasis, recent reports have suggest that not all immunosuppressive drugs necessarily promote HCC recurrence in transplant recipients. Sirolimus has emerged as a new, potent immunosuppressive agent which unlike other immunosuppressants [cyclosporine (CsA), tacrolimus (FK506), and azathioprine (AZA)] has potent antitumor activity in vitro and in vivo. The immunosuppressive and antitumor effects of sirolimus share a common mechanism of action. Sirolimus inhibits the mammalian target of sirolimus (mTOR), which prevents acute graft rejection mediated by interleukin-2 and could block other cytokine signal transduction, thus directly inhibits tumor cell proliferation and angiogenesis. And the most important is that the antitumor activity of SRL has been shown at the same concentrations as maintenance target levels in posttransplant patients.

Thus, it seems reasonable to speculate that sirolimus could simultaneously contribute to inhibition of tumor recurrence and preventing of rejection in OLT for patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

* The major organ (liver,heart, lung and kidney) function after OLT was normal.
* Pathologically proved HCC before randomisation .
* Tumor exceeding the Milan criteria (one nodule ≤5 cm or 2-3 nodules all <3 cm, without macroscopic vascular invasion and extrahepatic spreading).
* Signed, written informed consent.

Exclusion Criteria:

* Extrahepatic metastasis, nodal involvement, perioperative deaths (within 30 days after operation), and tumor thrombi in the proximal main trunk of the portal vein and / or vena cava
* History of cardiac disease.
* Active clinically serious infection (>grade 2 Nation Cancer Institute NCI-CTCAE version 3.0).
* Known history of human immunodeficiency virus (HIV) infection.
* Any condition that is unstable or which could jeopardize the safety of the patient and his / her compliance in the study.
* Pregnant or breast-feeding patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2007-08; Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3-,5-year

SECONDARY OUTCOMES:
overall survival | 3-,5-year

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD, Study Director — Liver Cancer Institute and Zhongshan Hospital, Fudan University, 200032, Shanghai, China.
Locations (1):
- Liver Cancer Institute and Zhongshan Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Derived] Treiber G. mTOR inhibitors for hepatocellular cancer: a forward-moving target. Expert Rev Anticancer Ther. 2009 Feb;9(2):247-61. doi: 10.1586/14737140.9.2.247. PMID 19192962